CLINICAL TRIAL: NCT05667714
Title: A Randomized, Single-blind, Placebo-controlled Clinical Trial to Evaluate the Efficacy and Safety of Anti-COVID-19 Antibody SA58 Nasal Spray, Among Close Contact With COVID-19 People
Brief Title: Efficacy and Safety of SA58 Nasal Spray in Close Contact With COVID-19 People
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sinovac Life Sciences Co., Ltd. (Industry)
Collaborators: Beijing Ditan Hospital (Other)
Responsible Party: Sponsor
Organization: Sinovac Biotech Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PRO-SA58-0002
Record Dates: First submitted 2022-12-13; First posted 2022-12-29 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2022-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental Group A（ non-continuous exposure to COVID-19） (Experimental): 1725 participants who were non-continuous exposure to COVID-19 received nasal spray every 3 hours,about 5-6 times/day.
  Interventions: Drug: SA58 Nasal Spray
- Control Group A（ non-continuous exposure to COVID-19） (Placebo Comparator): 575 participants who were non-continuous exposure to COVID-19 received nasal spray every 3 hours,about 5-6 times/day .
  Interventions: Drug: Placebo
- Experimental Group B (continuous exposure to COVID-19) (Experimental): 400 participants who were continuous exposure to COVID-19 received nasal spray every 3 hours,about 5-6 times/day.
  Interventions: Drug: SA58 Nasal Spray
- Control Group B(continuous exposure to COVID-19) (Placebo Comparator): 200 participants who were continuous exposure to COVID-19 received nasal spray every 3 hours,about 5-6 times/day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SA58 Nasal Spray — SA58 nasal spray , provided by Sinovac Life Sciences Co. , Ltd. mainly consists of neutralizing antibody of COVID-19, with 5 mg neutralizing antibody of COVID-19 per ml, 20 sprays per bottle.
  Arms: Experimental Group A（ non-continuous exposure to COVID-19）; Experimental Group B (continuous exposure to COVID-19)
Drug: Placebo — Placebo was provided by Sinovac Life Sciences Co. , Ltd.
  Arms: Control Group A（ non-continuous exposure to COVID-19）; Control Group B(continuous exposure to COVID-19)

SUMMARY:
This is a randomized, single-blind, placebo-controlled clinical trial to evaluate the efficacy and safety of SA58 nasal spray in close contact with COVID-19 people.

DETAILED DESCRIPTION:
This study is a randomized, single-blind, placebo-controlled clinical trial in close contacts to COVID-19. The investigational drug was manufactured by Sinovac Life Sciences Co. , Ltd.The purpose of this study is to estimate the efficacy and safety of SA58 nasal spray in close contacts to COVID-19. A total of 2900 subjects were planned to be enrolled,including 2300 subjects who were non-continuous exposed to COVID-19 in group A,600 subjects who were continuous exposed to COVID-19 in group B. All subjects started medication on the day of enrollment. During the medication period, the subjects were given nasal spray once every 3 hours,about 5-6 times a day.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 years and above on the day of enrollment;
* Had recent contact with an infected person, and the time of PCR sampling from a positive infected person, or the time of first contact with a positive infected person should not exceed 72 hours;
* The subjects can understand and voluntarily sign the informed consent form;

Exclusion Criteria:

* Previous history of severe allergy or sensitivity to inhalation allergens;
* Women are breastfeeding, pregnant, or planning to become pregnant during the study period;
* Participated in clinical trials of SARS-CoV-2 neutralizing antibody injections within 180 days prior to screening or clinical trials of other drugs within 4 weeks prior to screening;
* Subjects unable to cooperate with nasal spray inhalation;
* Body temperature at baseline (Day 0)>37.0℃;
* Had a severe neurological disorder (epilepsy, convulsions or convulsions) or psychosis, and have a family history of psychosis;
* The researchers determined that the subjects had a serious chronic medical condition that could interfere with the conduct or completion of the study;
* According to the investigator's judgment, the subject has any other factors that are not suitable for participating in the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2900 (Estimated)
Dates: Start 2022-11-26 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of symptomatic COVID-19 cases | Up to 30 days(during case surveillance period)
  Incidence of symptomatic COVID-19 cases confirmed by RT-PCR during case surveillance period

SECONDARY OUTCOMES:
Incidence of symptomatic COVID-19 cases confirmed by RT-PCR in subjects stratified by different Ct values at the time of diagnosis of primary cases(≤30, >30) | Up to 30 days (during case surveillance period)
  Incidence of symptomatic COVID-19 cases confirmed by RT-PCR when groups were stratified according to different Ct values at the time of diagnosis of primary cases(≤30, >30) during case surveillance period.
Incidence of symptomatic COVID-19 cases confirmed by RT-PCR in subjects stratified by actual dosing interval | Up to 30 days (during case surveillance period)
  Incidence of symptomatic COVID-19 cases confirmed by RT-PCR in subjects stratified by actual dosing interval during case surveillance period
The infection rate of asymptomatic COVID-19 infected people confirmed by RT-PCR | Up to 30 days (during case surveillance period)
  The infection rate of asymptomatic COVID-19 infected people confirmed by RT-PCR during the case surveillance period.
The incidence rate of symptomatic COVID-19 cases (mild, normal, severe and critical) | Up to 30 days (during case surveillance period)
  The incidence rate of symptomatic COVID-19 cases (mild, normal, severe and critical)during the case surveillance period.
The peak Ct value | Up to 30 days (during case surveillance period)
  The peak Ct value during the period of case surveillance
The number of days of infection | Up to 30 days (during case surveillance period)
  The number of days of infection during the period of case surveillance.

CONTACTS AND LOCATIONS:
Overall Officials: Ronghua Jin, Principal Investigator — Beijing Ditan Hospital
Locations (1):
- Beijing Ditan Hospital, Capital Medical University, Beijing, China